CLINICAL TRIAL: NCT03329053
Title: A Randomized Controlled Trial to Evaluate Utilization of Physical Activity Recommendations Among Patients of Cardiovascular Healthcare Centres in Eastern Slovakia: Study Design and Rationale of the AWATAR Study
Brief Title: Utilization of Physical Activity Recommendations Among Patients of Cardiovascular Healthcare Centres in Eastern Slovakia
Acronym: AWATAR
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study research team disintegration
Sponsor: Pavol Jozef Safarik University (Other)
Collaborators: University of Groningen (Other)
Responsible Party: Principal Investigator, Aurel Zelko, Institute of Physical Education and Sport, Pavol Jozef Safarik University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PJSU-1/0825/17
Record Dates: First submitted 2017-10-24; First posted 2017-11-01 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Cardiovascular Diseases
Keywords: exercise prescription; digital exercise prescription tool
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Equipment and Supplies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Patients randomized into the experimental group will undergo behavioural counselling. During the 30-minute long consultation patients will receive standard, usual-cardio-care lifestyle, hypertension and cardiovascular instructions, except recommendations for physical activities. This domain will be consulted exclusively through the digital training and decision support system EXPERT tool.
  Interventions: Behavioral: The EAPC Exercise Prescription (EXPERT) Tool
- Control group (Active Comparator): Patients randomized into the control group will receive standard, usual-cardio-care lifestyle, hypertension and cardiovascular instructions, also in the domain of recommendations for physical activities.
  Interventions: Behavioral: Standard Cardio-Care Lifestyle Counselling

INTERVENTIONS:
Behavioral: The EAPC Exercise Prescription (EXPERT) Tool — During the 30-minute long consultation subjects will receive standard, usual-cardio-care lifestyle, hypertension and cardiovascular instructions, except recommendations for physical activities. This domain will be consulted exclusively through the digital training and decision support tool.
  The EXPERT tool is an interactive digital training and decision support system for optimized exercise prescription in cardiovascular disease patients. The EXPERT tool was designed to provide optimized exercise prescription based on detailed overview of patient´s diagnosis, prognostics, complications and medication.
  Arms: Experimental group
Behavioral: Standard Cardio-Care Lifestyle Counselling — During the 30-minute long consultation subjects will receive standard, usual-cardio-care lifestyle, hypertension and cardiovascular instructions also in the domain of recommendations for physical activities. The exercise prescription process during consultation will be constructed in accordance with published guidelines and recommendations for secondary prevention of cardiovascular diseases.
  Arms: Control group

SUMMARY:
The aims of this trial are:

(A) to determine and compare the indices of exercise recommendations compliance after exercise prescription according to digital training and decision support system as compared to exercise prescription following the standard informative procedure among patients with cardiovascular disease.

(B) to determine whether health literacy moderates effect of exercise prescription according to digital training and decision support system on the indices of exercise recommendations compliance among patients with cardiovascular disease.

DETAILED DESCRIPTION:
The trial will compare the utilization of physical activity recommendation between the standard lifestyle informative procedure and the digital training and decision system informative procedure.

We hypothesize that a higher rate of compliance between seven-day exercise report and physical activity recommendations will be observed in the experimental group compared with three-months waiting group.

The goal is to recruit patients with a stable diagnosis, clinically defined as sufficiently healthy to participate in an optimized (safe and monitored) exercise programme. Based on the experience with similar projects completed on Cardiovascular Health Centres (CHC) expected attrition rate is 25%. Such a value and 400 participants as a target recruitment number still allows to keep 150 participants in both groups and a power of 80% to detect the differences between groups and across the time at an α level of 0,05 (two-tailed).

The trial will be supervised by a Data Safety and Monitoring Board consisting of one independent, internationally recognized clinical researcher, one representative (cardiologist) from each cooperating Cardiovascular Healthcare Centre as an advisor and experts in health psychology, exercise psychology, trial management and exercise physiology. The Board will be the policy and decision-making authority of the trial.

ELIGIBILITY:
Inclusion Criteria:

* receive information about perceived health benefits and risks connected with participation in the study based on disease severity from the treating cardiologist about participation in the study,
* willingness to accept randomization and participation in the assessment procedures,
* at recruitment moment, medical record of one or more below-listed cardiovascular diagnosis: coronary artery disease, coronary artery bypass graft surgery, or endoscopic traumatic coronary artery bypass graft surgery, compensated heart failure, cardiomyopathy, intermittent claudication, implantable cardioverter defibrillator or pacemaker, ventricular assist devices, heart transplantation, valve disease or surgery, congenital heart disease and non-severe pulmonary hypertension.

Exclusion Criteria:

* include the presence of below-listed specific cardiovascular conditions, significantly increasing risks of sudden cardiovascular events, also identified as potential contraindications of physical activity on cardiovascular patients: uncontrolled hypertension, decompensated heart failure, severe and symptomatic aortic stenosis, uncontrolled arrhythmia, severe pulmonary hypertension, acute coronary syndromes, acute myocarditis, endocarditis, or pericarditis, aortic dissection, Marfan syndrome or presence of malignancy (active cancer) or life-treating disease, bed-ridden status, participation or plan to participate in other study during trial execution or plan to move during the trial execution.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-02-23 (Actual); Primary Completion 2020-02-23 (Actual); Study Completion 2020-02-23 (Estimated)

PRIMARY OUTCOMES:
Change in exercise recommendations compliance at three months | Before the intervention and 1-5 days after three months follow up
  Compliance will be determined as agreement between indices of exercise prescription delivered by EXPERT tool and self-reported indices of exercise performed in monitoring periods (1 year and 7 days period).

SECONDARY OUTCOMES:
Change in body weight at three months | Before the intervention and 1-5 days after three months follow up
  Assessment of body weight with use of calibrated electronic scale (weight in kilograms).
Change in body height at three months | Before the intervention and 1-5 days after three months follow up
  Assessment of body height with use of stadiometer (height in centimetres).
Change in Body Mass Index at three months | Before the intervention and 1-5 days after three months follow up
  Calculation of Body Mass Index based on patient's body weight and body height (in meters). Body Mass Index will be calculated as body weight in kilograms divided by body height in meters squared.
Change in leisure time physical activities at three months | Before the intervention and 1-5 days after three months follow up
  To measure the prevalence of physical activities unqualified as sport-related or performance-oriented exercises we will measure leisure time behaviours of participants via International Physical Activity Questionnaire - Short Form (IPAQ-SF).
Change in clinical data at three months | Before the intervention and 1-5 days after three months follow up
  Clinical data will included a list of actual patient's cardiovascular disease, cardiovascular risk factors, other chronic non-cardiovascular co-morbidities, patient´s medication (type of medication), systolic and diastolic blood pressure (mmHg), blood total and low-density lipoprotein cholesterol concentration (mmol/l), fasting glycaemia (mmol/l), resting, and known patient´s adverse events registered during exercise testing.
Change in health literacy at three months | Before the intervention and 1-5 days after three months follow up
  The Health literacy level will be assessed using The Health Literacy Questionnaire (HLQ). This questionnaire comprises nine domains to provide a detailed profile of health literacy of populations, groups or patients of interest. The HLQ is divided into two parts which differ in response categories. Part 1 (domains 1-5) has 4 response categories rating the extent of agreement from 1 to 4. Part 2 (domains 6-9) has 5 response categories rating the level of difficulty from cannot do or always difficult (1), to always easy (5). Each domain was scored as the average of the item scores. The score ranges from 1 to 4 or 1 to 5 respectively, a higher score indicating higher level of health literacy.

CONTACTS AND LOCATIONS:
Overall Officials: Alena Bukova, PhD., Study Chair — Institute of Physical Education and Sport, Pavol Jozef Safarik University
Locations (1):
- Cardiology and Internal Medicine Ambulance, Košice, Slovakia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hansen D, Dendale P, Coninx K, Vanhees L, Piepoli MF, Niebauer J, Cornelissen V, Pedretti R, Geurts E, Ruiz GR, Corra U, Schmid JP, Greco E, Davos CH, Edelmann F, Abreu A, Rauch B, Ambrosetti M, Braga SS, Barna O, Beckers P, Bussotti M, Fagard R, Faggiano P, Garcia-Porrero E, Kouidi E, Lamotte M, Neunhauserer D, Reibis R, Spruit MA, Stettler C, Takken T, Tonoli C, Vigorito C, Voller H, Doherty P. The European Association of Preventive Cardiology Exercise Prescription in Everyday Practice and Rehabilitative Training (EXPERT) tool: A digital training and decision support system for optimized exercise prescription in cardiovascular disease. Concept, definitions and construction methodology. Eur J Prev Cardiol. 2017 Jul;24(10):1017-1031. doi: 10.1177/2047487317702042. Epub 2017 Apr 18. PMID 28420250
- [Derived] Zelko A, Bukova A, Kolarcik P, Bakalar P, Majercak I, Potocnikova J, Reijneveld SA, van Dijk JP. A randomized controlled trial to evaluate utilization of physical activity recommendations among patients of cardiovascular healthcare centres in Eastern Slovakia: study design and rationale of the AWATAR study. BMC Public Health. 2018 Apr 4;18(1):454. doi: 10.1186/s12889-018-5349-1. PMID 29618329